CLINICAL TRIAL: NCT04011540
Title: The Use of Patient Electronic Communication in Psychiatric Evaluation and Treatment
Brief Title: Digital Data in Mental Health Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 831246
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms; Anxiety Generalized
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive a personalized digital data dashboards throughout the two-month study period.
  Interventions: Behavioral: Digital data
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Digital data — Receiving digital data prior to a scheduled mental health session
  Arms: Intervention

SUMMARY:
The Use of Patient Electronic Communication in Psychiatric Evaluation and Treatment intends to better understand how digital data, social media, and electronic communication can be used in mental health therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years of age
2. Primarily English speaking (for language analysis)
3. Willing to share at least one digital data source this includes Facebook, Google searches, YouTube searches, or screen time by downloading a free application (app) on their smartphone.
4. Regular activity viewing and posting on social media sites, defined as once a month posting
5. Has a mental or behavioral health provider and/or has a provider from the Philadelphia Society of Clinical Psychologists and currently enrolled in mental or behavioral therapy
6. Attends therapy at least once a month and intends to remain in therapy for the next three months
7. Willing to share dashboard with their behavioral health provider
8. Able to provide informed consent
9. Owns a smartphone
10. If the patient downloads an app, they are willing to download and keep an app on their phone for 3 months

Exclusion Criteria:

1. Under 18 years of age
2. Non-English speaker
3. Patient is in severe distress, e.g. respiratory, physical, or emotional distress
4. Patient is intoxicated, unconscious, or unable to appropriately respond to questions
5. Not currently enrolled in mental therapy
6. Not expected to remain in mental therapy for the next three months
7. Not a regular social media poster, or does not use Facebook and/or Instagram and/or not willing to share
8. Unwilling to share social media summary dashboard with behavioral health provider
9. Patient with diagnosed psychosis
10. Does not own a smartphone
11. Unwilling to download and keep an app on their phone for 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine behavioral and mental health clinics, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 57 | 58
Completed | 48 | 52
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (9.9) | 32.2 (11.2) | 31.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 49 | 54 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 48 | 50 | 98
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life (HRQoL), RAND 36-Item Health Survey Changed Value (Baseline to 2 Months)
Description: The RAND 36-Item Health Survey is a set of generic, coherent, and easily administered health-related quality of life (HRQoL) measures. It explores eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each item is scored on a 0 to 100 range. The lowest and highest possible scores are 0 and 100, respectively. A high score defines a more favorable health state (better outcome).
Time Frame: 2 months
Population: Changes value from baseline to 2 months. Note: the number of participants analyzed differs from total enrolled due to participants not completing the follow-up survey.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 48 | 52
score on a scale | -0.89 [-5.55 to 3.77] | -1.85 [-5.73 to 2.04]

2. Secondary Outcome: Depressive Symptoms, Patient Health Questionnaire-8 (PHQ-8) Change Value
Description: Patient health questionnaire-8 (PHQ-8) (Kroenke, Spitzer, & Williams, 2001) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-8 incorporates DSM-IV depression diagnostic criteria. Each question is rated on a scale of 0 to 3, minimum score is 0 and maximum score is 24. A total of 8 questions are administered. Lower scores indicate minimal depression (better outcome) and higher scores indicate severe depression (worse outcome).
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 47 | 52
score on a scale | -1.20 [-2.31 to -0.08] | -0.44 [-1.65 to 0.77]

3. Secondary Outcome: Anxiety Symptoms, Generalized Anxiety Disorder-7 (GAD-7) Change Value
Description: GAD-7 is a 7-item anxiety scale. It has good reliability, as well as criterion, construct, factorial, and procedural validity. Each item is rated according to the frequency of the described problem. The responses are scored as follows: 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day with a maximum score of 21 Scores are interpreted as 5 to 9, mild anxiety; 10 to 14, moderate anxiety; and 15 and above, severe anxiety. Lower scores represent mild anxiety (better outcome) while higher scores represent severe anxiety (worse outcome).
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 47 | 52
score on a scale | -0.90 [-2.10 to 0.30] | -1.14 [-2.38 to 0.10]

4. Secondary Outcome: Therapeutic Relationship, Working Alliance Inventory (WAI) Change Value
Description: Working Alliance Inventory (WAI) (Horvath and Greenberg 1986) is used to measure the service user-psychiatrist relationship from the service user perspective. The Working Alliance Inventory-Short Version (WAI-S) is based upon Bordins three-factor conceptualization of the provider and client relationship: collaboration on tasks, collaboration on goals and the bond between the client and therapist. Participants rate items on a 5-point Likert scale anchored at each end with 'rarely or never' (1) and 'always' (5). The total score is simply the sum of all the scores with the appropriate negative items reversed prior to summing. The total score ranges from 5 to 20. Higher scores indicate a better therapeutic alliance (better outcome). Higher positive mean change score represents 'worsened' alliance, whereas negative mean change score represents 'improved' alliance.
Time Frame: 2 months
Population: Mean change values from baseline to 2 months. Note: the number of participants analyzed differs from total enrolled due to participants not completing the follow-up survey.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 47 | 52
score on a scale | 0.36 [-1.52 to 2.25] | -0.65 [-2.26 to 0.95]

ADVERSE EVENTS:
Time Frame: Not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT04011540/Prot_SAP_000.pdf